CLINICAL TRIAL: NCT04919551
Title: A Clinical Trial to Evaluate the Effect of Food on PK and PD of Vicagrel Capsules in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VCP1-Ⅰ-05
Record Dates: First submitted 2021-06-08; First posted 2021-06-09 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — methyl 2-(2-acetoxy-6,7-dihydrothieno(3,2-c)pyridin-5(4H)-yl)-2-(2-chlorophenyl)acetate

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, open-label, single-dose, fasted/high-fat meal/low-fat meal, 3-cycle, 3-way crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- KGD (Experimental): Oral administration after fasting/high-fat meal/low-fat meal
  Interventions: Drug: vicagrel
- GDK (Experimental): Oral administration after high-fat meal/low-fat meal/fasting
  Interventions: Drug: vicagrel
- DKG (Experimental): Oral administration after low-fat meal/fasting/high-fat meal
  Interventions: Drug: vicagrel

INTERVENTIONS:
Drug: vicagrel — Oral administration after fasting/high-fat meal/low-fat meal

SUMMARY:
This clinical study will adopt a randomized, open-label, single-dose, 3-cycle, 3-way crossover design to explore the PK and PD profiles of a single oral dose of vicagrel capsules under fasted and fed conditions in health subjects.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signing of informed consent before the trial, and full understanding of the experimental content, process and possible ARs;
* Able to complete the study according to the protocol;
* Subjects (and their partners) are willing to take effective contraceptive measures from screening to 6 month after the last dose of the IMPs. See Appendix 5 for specific contraceptive measures;
* Male and female subjects aged 18 to 45 years (inclusive);
* Male weight ≥50 kg, female weight ≥ 45 kg. Body mass index (BMI) = body weight (kg) / height2 (m2). BMI ranging from 18 to 28 kg/m2 (including critical values);
* Physical examination and vital signs are normal or abnormal without clinical significance.

Exclusion Criteria:

* More than 5 cigarettes per day on average 3 months before the trial;
* Allergic constitution (allergic to multiple drugs and foods), or known to be possibly allergic to drugs of the same class of the IMP or highly sensitive to clopidogrel;
* History of alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine); history of drug abuse or use of hard drug within the past five years;
* Blood donation or massive blood loss (>450 mL) within 3 months before screening;
* Presence of dysphagia or history of any gastrointestinal and hepatic, renal disease (whether cured or not) or history of surgery that affects absorption or excretion of the IMP within 6 months prior to screening;
* With any disease that increases the risk of bleeding, such as acute gastritis, stomach and duodenal ulcers, or history of abnormal bleeding (e.g. bleeding time prolonged after tooth extraction);
* The subject or his or her immediate family member has a family history of coagulation or haemorrhagic disorders (such as haemophilia)/symptoms (such as hematemesis, melena, severe or recurrent epistaxis, coughing blood (hemoptysis), obvious hematuria or intracranial hemorrhage), or suspected vascular malformation, such as aneurysm or early-onset stroke;
* Took potent inhibitors and/or inducers of CYP enzymes (CYP1A2, 2A6, 2C8, 2C19, 3A4 and 3A5) within 28 days prior to the first dose. Potent inhibitors of CYP enzymes include ciprofloxacin, clopidogrel, itraconazole, ketoconazole, ritonavir, troleandomycin, etc.. Potent inducers of CYP enzymes include rifampicin, carbamazepine, phenytoin sodium, St. John's wort, etc.. See Appendix 6 for details;
* Took any prescription, non-prescription, any vitamin or herbal drugs within 14 days before the first dose;
* Had foods that affect CYP3A4 metabolism within 2 weeks prior to the first dose, such as grapefruit or grapefruit-containing beverages, or had intense physical exercise (e.g. strength training, aerobic training, and playing football) within 7 days prior to the first dose, or other factors affecting drug absorption, distribution, metabolism, excretion, etc.;
* Recently there have been major changes in diet or exercise habits;
* Participated in a another clinical study within 3 months prior to screening (a subject may be enrolled if he/she withdraws from the study prior to treatment, i.e., the subject is not randomized or doesn't receive treatment);
* Failure to tolerate high-fat meals (two boiled eggs, one slice of toast with butter and bacon, a box of French fries, a glass of whole milk);
* 12-lead ECG abnormalities have clinical significance;
* Female subjects who are in lactation or positive for serum pregnancy test in the screening period or during the trial;
* Clinical laboratory abnormalities have clinical significance or other clinically significant diseases before screening (including but not limited to gastrointestinal, kidney, liver, nerve, blood, endocrine, tumor, and lung, immune, mental or cardiovascular and cerebrovascular diseases);
* Positive for viral hepatitis (including hepatitis B and C), HIV antibody and treponema pallidum antibody during screening;
* Any acute diseases or concomitant medicines from screening period to before taking the IMPs;
* Took chocolate, any food or drink with caffeine or xanthine within 24 hours before the first dose;
* Took any alcoholic product or alcohol breath test is positive within 24 hours before the first dose;
* Urine drug screening positive;
* The investigator believes that there are other factors that are not suitable for participating in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
AUC | 48 hours
  Area Under the Curve From Time Zero to Last Quantifiable Concentration
Cmax | 48 hours
  Peak concentration

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China